CLINICAL TRIAL: NCT04460950
Title: A Retrospective and Prospective Multicentre Observational Study for the Evaluation of Incidence of Familial AML/MDSs in Patients With Myeloid Neoplasms (AML/MDS)
Brief Title: Observational Study for the Evaluation of Incidence of Familial AML/MDSs in Patients With Myeloid Neoplasms
Status: Recruiting | Type: Observational
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: AML2120
Record Dates: First submitted 2020-06-25; First posted 2020-07-08 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Acute Myeloid Leukemia; Familial Acute Myeloid Leukemia; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
Observational study aimed at evaluating the incidence of familial AML/MDSs in patients with de novo MDSs or AML with almost one relative affected by hematologic neoplasms and/or other cancers at young age (< 40 years)

DETAILED DESCRIPTION:
This is a multicenter, retrospective and prospective, observational study aims to collect clinical information on patients with familial AML/MDSs from January 2014 to December 2022. No intervention is expected.

The purpose of this study is to identify and characterize the patients with familial MDSs or AML (i.e. with relatives affected by hematologic neoplasms and/or other cancers at young age (< 40 years)) or presence of signs, symptoms or laboratory tests compatible with one of the known syndromes with germinal susceptibility to AML/MDSs.

In order to estimate the incidence of familial AML/MDSs, a survey will be sent every year to all participating sites to collect only the number of the all diagnosis of AML/MDS. All patients will be followed until December 2023 in order to have at least 1 year of observation.

ELIGIBILITY:
Inclusion Criteria:

* Patient age > 18 years old
* Diagnosis of AML or MDSs from January 2014 to December 2022
* Suspected familiarity for myeloid neoplasm: at least one family member of first or second degree affected by myeloid neoplasm or other hematological malignancy, or by solid tumors with onset at age < 40 years or presence of signs, symptoms or laboratory tests compatible with one of the known syndromes with germinal susceptibility to AML/MDSs
* Signed written informed consent according to ICH/EU/GCP and national local laws.

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnoses with AML and MDSs from January 2014 to December 2022 will be registered. Study population will include patients with MDSs or AML with at least one family member of first or second degree affected by myeloid neoplasm or other hematological malignancy, or by solid tumors with onset at age < 40 years.
Sampling Method: Non-Probability Sample
Enrollment: 237 (Estimated)
Dates: Start 2020-12-16 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of familial AML/MDSs | at 1 year
  Evaluation of incidence of familial AML/MDSs in patients with de novo MDSs or AML with almost one relative affected by hematologic neoplasms and/or other cancers at young age (< 40 years). The incidence of familial AML/MDSs will be evaluated by means of number of diagnosis of familial AML/MDSs on the number of all diagnosis of AML/MDS between January 2014 and December 2022.

SECONDARY OUTCOMES:
Hematological characteristics of familial AML/MDSs | at 1 year
  Evaluation of hematological characteristics of patients with familial AML/MDS.
Distribution of familial hematologic neoplasms and/or other cancers | at 1 year
  Type and rate of familial hematologic neoplasms and/or other cancers
Incidence of transplantation | at 1 year
  Outcome of transplant in patients with familial AML/MDS
Survival Distribution | at 1 year
  Overall Survival (OS) and Progression Free Survival (PFS)
Standardized Mortality Ratio (SMR) | at 1 year
  SMR to compare the survival risk in patients with familial AML/MDS with the risk in the Italian general population

CONTACTS AND LOCATIONS:
Locations (27):
- Italy (27):
  - Aon Ss. Antonio E Biagio E C. Arrigo - Alessandria - Soc Ematologia, Alessandria
  - Aou Ospedali Riuniti "Umberto I - G.M. Lancisi - G. Salesi"- Ancona - Sod Clinica Ematologica, Ancona
  - Ao Di Rilievo Nazionale E Di Alta Specialità "San Giuseppe Moscati" - Avellino - Uoc Ematologia Con Unità Di Trapianto, Avellino
  - Asl Caserta, Presidio Ospedaliero S.G.Moscati - Aversa - Uo Oncoematologia, Aversa
  - Aou Di Bologna - Policlinico S. Orsola-Malpighi - Uoc Ematologia, Bologna
  - Asst Degli Spedali Civili Di Brescia - Ssvd Centro Trapianti Midollo Per Adulti - Cattedra Di Ematologia, Brescia
  - Asst Degli Spedali Civili Di Brescia - Uo Ematologia, Brescia
  - Ao Brotzu, Presidio Ospedaliero A. Businco - Cagliari - Sc Ematologia E Ctmo, Cagliari
  - Aou Ospedali Riuniti - Foggia - Uoc Ematologia, Foggia
  - Asl Lecce, Ospedale 'V. Fazzi' - Uo Ematologia, Lecce
  - Ao Ospedali Riuniti "Papardo Piemonte" - Po Papardo - Messina - Sc Ematologia, Messina
  - Asst Grande Ospedale Metropolitano Niguarda - Milano - Sc Ematologia, Milan
  - Fondazione Irccs Ca' Granda, Ospedale Maggiore Policlinico - Milano - Ematologia - Padiglione Marcora, Milan
  - Aou San Luigi Gonzaga - Orbassano - Scdu Ematologia Generale E Oncoematologia, Orbassano
  - Asl Salerno, Presidio Ospedaliero Tortora Pagani - Ematologia, Pagani
  - Aou Policlinico P. Giaccone - Palermo - Uo Ematologia, Palermo
  - Aou Di Parma - Sc Ematologia E Centro Trapianti Midollo Osseo, Parma
  - Ao Di Perugia, Ospedale S. Maria Della Misericordia - Ematologia E Trapianto Midollo Osseo, Perugia
  - Aou Pisana - Uo Ematologia Universitaria, Pisa
  - Ausl Di Reggio Emilia - Arcispedale Santa Maria Nuova, Irccs - Sc Ematologia, Reggio Emilia
  - Ausl Della Romagna, Ospedale "Infermi" - Rimini - Uo Ematologia, Rimini
  - Asl Roma 2, Ospedale S. Eugenio- Ospedale S.Eugenio - Uoc Ematologia, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli Irccs - Roma - Area Ematologica, Roma
  - Ente Ecclesiastico Casa Sollievo Della Sofferenza - San Giovanni Rotondo - Ematologia, San Giovanni Rotondo
  - Aou Di Sassari - Cliniche Universitarie - Stabilimento Cliniche Di San Pietro - Uoc Ematologia, Sassari
  - Aou Città Della Salute E Della Scienza, Ospedale S. Giovanni Battista Molinette - Torino - Sc Ematologia - Università Degli Studi Di Torino, Torino
  - Asui Di Udine - Presidio Ospedaliero "Santa Maria Della Misericordia" - Clinica Ematologica, Udine